CLINICAL TRIAL: NCT03000309
Title: Use of Apremilast in Patients Who Are Dissatisfied With Stable Maintenance Topical Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APR-2015
Record Dates: First submitted 2016-12-15; First posted 2016-12-22 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apremilast (Other): Apremilast, 30 mg. tablets, two times a day for 16 weeks
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast
  Other Names: Otezla

SUMMARY:
Sixteen week open label study of apremilast in combination with topical steroids with a four week safety follow up visit.

DETAILED DESCRIPTION:
This is an open label, 16 week study of apremilast in combination with topical corticosteroids (TCS). Twenty qualified subjects will be enrolled. Visits will consist of Baseline, 8 week, 16 week and a 20 week safety follow up after 4 weeks off treatment. Subjects will dose with apremilast as per label. Topical corticosteroids (TCS) will be used for up to Week 4 as per label and then will be used on an as needed basis until Week 16. Assessments will include Static Physicians Global Assessment (sPGA), Psoriasis Area Severity Index (PASI), Psoriatic Body Surface Area (BSA), Dermatology Life Quality Index (DLQI),Assessment of Pruritus, Patient Satisfaction questionnaire. and Patient Global Assessment (PtGA)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be in general good health as judged by investigator
* Female of childbearing potential (FCBP) must have a negative pregnancy test at screening and Baseline.
* FCBP must use an approved method of contraception as outlined in the protocol.
* Male subjects who engage in activity in which conception is possible must use barrier contraception as defined in the protocol.
* 18 years of age or older
* Understand and voluntarily sign the Informed Consent
* Able to adhere to study visit schedule
* Moderate plaque type psoriasis as define by a a PGA of 3
* BSA 0f 5-10% or a DLQI score of 7 or more
* History of uncontrolled plaque psoriasis after either stable dose of high potency topical steroids for 2 weeks or mid-potency steroids for 4 weeks within the last 6 months

Exclusion Criteria:

* Any clinically significant disease as determined by the investigator or major disease that is currently uncontrolled
* Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk
* Prior history of suicide attempt at any time in the subject's lifetime prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years
* Pregnant or breastfeeding, FCBP who are not willing to use acceptable birth control methods.
* Active substance abuse or a history of substance abuse within 6 months prior to screening.
* Malignancy or history of malignancy except fo treated (cured) basal cell or or squamous cell in situ skin carcinomas, treated (cured) cervical intraepithelial neoplasia or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years
* Has not completed the prescribed washout for restricted treatments
* Known or suspected allergy to investigational product
* Other types of psoriasis
* Prior history of depression
* Prior use of apremilast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H. Kircik, M.D., Principal Investigator — DermResearch PLLC
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Apremilast: Apremilast, 30 mg. tablets, two times a day for 16 weeks
  Apremilast
Period: Overall Study
Arm/Group | Apremilast
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Apremilast
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  black | 2
  white | 18
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Product of BSA (Body Surface Affected by Psoriasis) and sPGA (Static Physician Global Assessment) From Baseline to Week 16
Description: The area of body surface affected by psoriasis (BSA) will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. Static Physician Global Assessment (sPGA) of disease severity is measured by the Investigator on a 6-point scale wherein 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, 4=Severe, 5=Very Severe. The product of these values offers a more specific assessment of the severity of psoriasis. This product can yield a result between 0 (no disease) and 500 (most severe disease) By reporting the percent change as well as the absolute value change, the reader may be better able to appreciate the impact on disease severity of the medication under study.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 20
score on a scale | -9 (10)

2. Primary Outcome: Percent Change in Product of BSA and sPGA
Description: The area of body surface affected by psoriasis (BSA) will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. Static Physician Global Assessment (sPGA) is measured by the Investigator on a 6-point scale wherein 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, 4=Severe, 5=Very Severe. The product of these values offers a more specific assessment of the severity of psoriasis. This product can yield a result between 0(no disease) and 500 (most severe disease.) By reporting the percent change as well as the absolute value change, the reader may be better able to appreciate the impact on disease severity of the medication under study.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 20
percent change | -44 (52)

3. Secondary Outcome: Percent Change in Product of BSA and sPGA
Description: The area of body surface affected by psoriasis (BSA) will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. Static Physician Global Assessment (sPGA) is measured by the Investigator on a 6-point scale wherein 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, 4=Severe, 5=Very Severe. Th3 product of these values offers a more specific assessment of the severity of psoriasis. This product may yield a result between 0 (no disease) and 500 (most severe disease.)
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 20
percent change | -29 (36)

4. Secondary Outcome: Mean Change in DLQI
Description: The Dermatology Life Quality Index (DLQI) is a 10-question survey administered to subjects in order to ascertain the extent to which psoriasis has affected the patient's life in the week prior to completing the questionnaire. The score is a sum of the value of each answer wherein Very Much=3, A lot=2, A little=1 and Not at all=0. 0 is the lowest possible score and indicates no impact of disease on quality of life. 30 is the highest possible score and indicates the most negative impact of disease on quality of life.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 20
score on a scale | -6 (5)

5. Secondary Outcome: Mean Change in DLQI
Description: as for outcome 4
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 20
units on a scale | -7 (5)

6. Secondary Outcome: Mean Change in Pruritus Scores
Description: The Subject Assessments of pruritis is measured at screening, baseline, and weeks 4, 8 and 16. Each subject rates the severity of their itching over the last 24 hours on a 10-point scale from 0 (none) to 10 (unbearable)
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 20
units on a scale | -3 (2)

7. Secondary Outcome: Mean Change in Pruritus Scores
Description: as for outcome 6
Time Frame: Baseline to Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 20
units on a scale | -3 (3)

8. Secondary Outcome: Mean Change in BSA
Description: The area of body surface affected by psoriasis (BSA) will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. This will be assessed at screening, baseline, and weeks 4, 8 and 16
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: percentage of body surface area affected
Arm/Group | Apremilast
Number analyzed (Participants) | 20
percentage of body surface area affected | -1 (2)

9. Secondary Outcome: Mean Change in BSA
Description: as for outcome 8
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: percentage of body surface area affected
Arm/Group | Apremilast
Number analyzed (Participants) | 20
percentage of body surface area affected | -2 (3)

10. Secondary Outcome: Percent Change in BSA
Description: as for outcome 8
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 20
percent change | -19 (28)

11. Secondary Outcome: Percent Change in BSA
Description: as for outcome 8
Time Frame: Baseline to Week 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 20
percent change | -36 (49)

12. Secondary Outcome: Proportion of Patients Who Achieve PASI 50
Description: The Psoriasis Area Severity index (PASI) is performed at screening, baseline, and weeks 4, 8 and 16. This tool is used to measure the severity and extent of disease by combining the assessment of severity of lesions and the area affected into a single score in the range of 0 (no disease) to 72 (maximal disease.)
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 20
Participants | 3

13. Secondary Outcome: Proportion of Patients Who Achieve PASI 50
Description: as for outcome 12
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 20
Participants | 8

14. Secondary Outcome: Proportion of Patients Who Achieve PASI 75
Description: as for outcome 12
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 20
Participants | 0

15. Secondary Outcome: Proportion of Patients Who Achieve PASI 75
Description: as for outcome 12
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 20
Participants | 6

16. Secondary Outcome: % of Patients Achieving Clear or Almost Clear on the PtGA
Description: as for outcome 12
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 20
Participants | 10

17. Secondary Outcome: % of Patients Achieving Clear or Almost Clear on the PtGA
Description: as for outcome 12
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 20
Participants | 9

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Apremilast
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 17/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=20)
headache (General disorders) | 5 (5)
diarrhea (Gastrointestinal disorders) | 6 (6)
irritability (General disorders) | 1 (1)
upset stomach, unspecified (Gastrointestinal disorders) | 3 (3)
nausea (Gastrointestinal disorders) | 6 (6)
leg cramps (General disorders) | 1 (1)
upper respiratory infection (Infections and infestations) | 1 (1)
otitis externa (Infections and infestations) | 1 (1)
abdominal cramping (Gastrointestinal disorders) | 3 (3)
viral gastroenteritis (Gastrointestinal disorders) | 1 (1)
cyst left inner thigh (Skin and subcutaneous tissue disorders) | 1 (1)
abscess right hand (Skin and subcutaneous tissue disorders) | 1 (1)
heartburn (Gastrointestinal disorders) | 2 (2)
right flank pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT03000309/Prot_SAP_000.pdf